CLINICAL TRIAL: NCT00377637
Title: A Prospective, Randomized, Active Controlled, Parallel Group, Multi-center Trial to Assess the Efficacy and Safety of Mycophenolate Mofetil (MMF) in Inducing Response and Maintaining Remission in Subjects With Lupus Nephritis.
Brief Title: A Study of Mycophenolate Mofetil (CellCept) in Management of Patients With Lupus Nephritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Aspreva Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WX17801; NCT00121082 (obsolete NCT alias)
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-10

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Mycophenolic Acid; Cyclophosphamide; Azathioprine; Adrenal Cortex Hormones

ARMS (4):
- Induction Phase: Mycophenolate mofetil (Experimental): Participants received oral mycophenolate mofetil (MMF) 1.5 g twice a day and concomitant corticosteroids for the 24 weeks of the Induction Phase.
  Interventions: Drug: Mycophenolate mofetil (MMF); Drug: Corticosteroid
- Induction Phase: Cyclophosphamide (Active Comparator): Participants received monthly infusions of cyclophosphamide, 0.5 to 1.0 g per square meter of body surface area and concomitant treatment with corticosteroids for the 24 week Induction Phase.
  Interventions: Drug: Cyclophosphamide; Drug: Corticosteroid
- Maintenance Phase: Mycophenolate mofetil (Experimental): Participants received mycophenolate mofetil (MMF) 1.0 g orally twice a day, placebo to azathioprine orally once a day and corticosteroid for the 36 weeks Maintenance Phase.
  Interventions: Drug: Mycophenolate mofetil (MMF); Drug: Placebo to Azathioprine; Drug: Corticosteroid
- Maintenance Phase: Azathioprine (Active Comparator): Participants received azathioprine (AZA) 2 mg/kg/day orally once a day, placebo to mycophenolate mofetil orally twice a day and corticosteroid for the 36 weeks Maintenance Phase.
  Interventions: Drug: Azathioprine; Drug: Placebo to Mycophenolate mofetil; Drug: Corticosteroid

INTERVENTIONS:
Drug: Mycophenolate mofetil (MMF) — Supplied as 500 mg tablets taken orally twice a day (BID). Dose specific for each arm. Dosing started at 500 mg BID for the first week, increasing by 500 mg in subsequent weeks until the final target dose was reached.
  Other Names: CellCept
  Arms: Induction Phase: Mycophenolate mofetil; Maintenance Phase: Mycophenolate mofetil
Drug: Cyclophosphamide — Intravenous cyclophosphamide (IVC) was administered every four weeks (monthly) to a total of six infusions.
  Dosing was started at 0.75 g/m^2 of body surface area for the first month, with subsequent doses at 0.5-1.0 g/m^2. The target dose was 1.0 g/m^2, but doses were titrated by 0.25 g/m^2 increments to maintain nadir leukocyte count between 2500-4000/mm^3.
  Other Names: Endoxan®
  Arms: Induction Phase: Cyclophosphamide
Drug: Azathioprine — 2 mg/kg/day orally, provided as 50 mg capsules to be taken after meals.
  Other Names: Imuran®
  Arms: Maintenance Phase: Azathioprine
Drug: Placebo to Azathioprine — Placebo capsules matching Azathioprine taken orally once a day.
  Arms: Maintenance Phase: Mycophenolate mofetil
Drug: Placebo to Mycophenolate mofetil — Placebo tablets matching Mycophenolate mofetil taken orally twice daily.
  Arms: Maintenance Phase: Azathioprine
Drug: Corticosteroid — Oral prednisolone (or equivalent) starting at a dose of 0.75-1.0 mg/kg/day (maximum 60 mg/day) tapered to 10 mg/day.

SUMMARY:
This 2 arm study assessed the efficacy of Mycophenolate Mofetil (MMF; CellCept) compared to cyclophosphamide in inducing a response in patients with lupus nephritis, and the long term efficacy of MMF compared to azathioprine in maintaining remission and renal function. Patients were randomized to receive either MMF (1.5 g twice daily [bid]) or cyclophosphamide (0.5-1.0 g/m^2 in monthly pulses) in the induction phase. Those patients meeting criteria for response were re-randomized for entry into the maintenance phase, to receive either MMF (1 g bid) or azathioprine (2 mg/kg/day).

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, 12-75 years of age;
* diagnosis of systemic lupus erythematosus;
* kidney biopsy within 6 months of study, with histological diagnosis of lupus nephritis;
* laboratory evidence of active nephritis.

Exclusion Criteria:

* continuous dialysis starting >2 weeks before randomization into induction phase, and/or with an anticipated duration of >8 weeks;
* previous or planned kidney transplant;
* other clinically significant active medical conditions.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2005-07; Primary Completion 2007-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (97):
- United States (25):
  - Huntsville, Alabama
  - La Jolla, California
  - Los Angeles, California
  - San Francisco, California
  - San Leandro, California
  - Torrance, California
  - Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Columbia, Missouri
  - Brooklyn, New York
  - Lake Success, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - San Isidro
  - San Miguel de Tucumán
- Australia (5):
  - Adelaide
  - Camperdown
  - Melbourne
  - Parkville
  - Woodville
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- Brazil (3):
  - Rio de Janeiro
  - São Paulo
  - Sorocaba
- Canada (6):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- China (5):
  - Beijing
  - Guangdong
  - Guangzhou
  - Jiangsu
  - Shanghai
- Czechia (2):
  - Brno
  - Prague
- France (5):
  - Lille
  - Lyon
  - Nantes
  - Paris
  - Toulouse
- Germany (10):
  - Aachen
  - Bad Bramstedt
  - Berlin
  - Dresden
  - Düsseldorf
  - Erlangen
  - Hanover
  - Leipzig
  - München
  - Münster
- Greece (2):
  - Athens
  - Heraklion
- Hungary (3):
  - Debrecen
  - Pécs
  - Szeged
- Italy (5):
  - Brescia
  - Milan
  - Padua
  - Pisa
  - Udine
- Mexico (3):
  - Mexico City
  - Mérida
  - San Luis Potosí City
- Portugal (2):
  - Lisbon
  - Porto
- Spain (6):
  - Alicante
  - Barcelona
  - Madrid
  - Málaga
  - Santander
  - Seville
- United Kingdom (8):
  - Birmingham
  - Cambridge
  - Leeds
  - London
  - Manchester
  - Newcastle upon Tyne
  - Sheffield
  - Southampton

REFERENCES:
- [Derived] Sundel R, Solomons N, Lisk L; Aspreva Lupus Management Study (ALMS) Group. Efficacy of mycophenolate mofetil in adolescent patients with lupus nephritis: evidence from a two-phase, prospective randomized trial. Lupus. 2012 Nov;21(13):1433-43. doi: 10.1177/0961203312458466. Epub 2012 Aug 24. PMID 22922564
- [Derived] Dooley MA, Jayne D, Ginzler EM, Isenberg D, Olsen NJ, Wofsy D, Eitner F, Appel GB, Contreras G, Lisk L, Solomons N; ALMS Group. Mycophenolate versus azathioprine as maintenance therapy for lupus nephritis. N Engl J Med. 2011 Nov 17;365(20):1886-95. doi: 10.1056/NEJMoa1014460. PMID 22087680
- [Derived] Dall'Era M, Stone D, Levesque V, Cisternas M, Wofsy D. Identification of biomarkers that predict response to treatment of lupus nephritis with mycophenolate mofetil or pulse cyclophosphamide. Arthritis Care Res (Hoboken). 2011 Mar;63(3):351-7. doi: 10.1002/acr.20397. Epub 2010 Nov 15. PMID 21080348
- [Derived] Ginzler EM, Wofsy D, Isenberg D, Gordon C, Lisk L, Dooley MA; ALMS Group. Nonrenal disease activity following mycophenolate mofetil or intravenous cyclophosphamide as induction treatment for lupus nephritis: findings in a multicenter, prospective, randomized, open-label, parallel-group clinical trial. Arthritis Rheum. 2010 Jan;62(1):211-21. doi: 10.1002/art.25052. PMID 20039429
- [Derived] Isenberg D, Appel GB, Contreras G, Dooley MA, Ginzler EM, Jayne D, Sanchez-Guerrero J, Wofsy D, Yu X, Solomons N. Influence of race/ethnicity on response to lupus nephritis treatment: the ALMS study. Rheumatology (Oxford). 2010 Jan;49(1):128-40. doi: 10.1093/rheumatology/kep346. Epub 2009 Nov 20. PMID 19933596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The induction phase was a prospective, randomized, open-label, active controlled, parallel group, international multicenter, 2-arm comparison study of MMF versus IVC in inducing a response in patients with Lupus nephritis. Responders in the induction phase were re-randomized into a double-blind, double-dummy, active controlled Maintenance Phase.
Groups:
- Induction Phase: Cyclophosphamide: Participants received monthly intravenous infusions of cyclophosphamide, 0.5 to 1.0 g per square meter of body surface area and concomitant treatment with corticosteroids for the 24 week Induction Phase.
- Induction Phase: Mycophenolate Mofetil: Participants received oral mycophenolate mofetil (MMF) 1.5 g twice a day and concomitant corticosteroids for the 24-weeks of the Induction Phase.
- Maintenance Phase: Mycophenolate Mofetil: Participants who responded to Induction Phase treatment received mycophenolate mofetil (MMF) 1.0 g orally twice a day, placebo to azathioprine orally once a day and corticosteroid for the 36 weeks Maintenance Phase.
- Maintenance Phase: Azathioprine: Participants who responded to Induction Phase treatment received azathioprine (AZA) 2 mg/kg/day orally once a day, placebo to mycophenolate mofetil orally twice a day and corticosteroid for the 36 weeks Maintenance Phase.
Period: Induction Phase
Arm/Group | Induction Phase: Cyclophosphamide | Induction Phase: Mycophenolate Mofetil | Maintenance Phase: Mycophenolate Mofetil | Maintenance Phase: Azathioprine
Started | 185 (Intent-To-Treat) | 185 (Intent-To-Treat) | 0 | 0
Safety Population | 180 | 184 | 0 | 0
Completed | 156 | 150 | 0 | 0
Not Completed | 29 | 35 | 0 | 0
Not completed — Adverse Event | 12 | 21 | 0 | 0
Not completed — Deterioration/serum creatinine | 2 | 0 | 0 | 0
Not completed — Dose reduction of MMF < 2 g/day for 14 d | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Death | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 6 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 0 | 0
Not completed — Sponsor decision | 1 | 2 | 0 | 0
Not completed — Non-Compliance | 1 | 0 | 0 | 0
Not completed — Reason for withdrawal is not noted | 2 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Induction Phase: Cyclophosphamide | Induction Phase: Mycophenolate Mofetil | Maintenance Phase: Mycophenolate Mofetil | Maintenance Phase: Azathioprine
Started | 0 | 0 | 116 | 111
Completed | 0 | 0 | 73 | 54
Not Completed | 0 | 0 | 43 | 57
Not completed — Adverse Event | 0 | 0 | 29 | 43
Not completed — Physician Decision | 0 | 0 | 5 | 4
Not completed — Lost to Follow-up | 0 | 0 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3
Not completed — Sponsor decision | 0 | 0 | 2 | 3
Not completed — Non-compliance | 0 | 0 | 1 | 1
Not completed — Study medication stopped > 14 days | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction Phase: Cyclophosphamide | Induction Phase: Mycophenolate Mofetil | Maintenance Phase: Mycophenolate Mofetil | Maintenance Phase: Azathioprine | Total
Number analyzed (Participants) | 185 | 185 | 116 | 111 | 597
Age, Customized [Mean (Standard Deviation); unit: years]
  Induction Phase | 31.3 (10.25) | 32.4 (11.7) | NA (NA) — Did not participate in the Induction Phase. Please see Maintenance Phase. | NA (NA) — Did not participate in the Induction Phase. Please see Maintenance Phase. | 31.9 (10.72)
  Maintenance Phase | NA (NA) — Did not participate in the Maintenance Phase. Please see Induction Phase. | NA (NA) — Did not participate in the Maintenance Phase. Please see Induction Phase. | 31.8 (10.59) | 31.0 (10.77) | 31.4 (10.65)
Sex/Gender, Customized [Number; unit: Participants]
  Induction Phase - Female | 156 | 157 | 0 | 0 | 313
  Induction Phase - Male | 29 | 28 | 0 | 0 | 57
  Maintenance Phase - Female | 0 | 0 | 99 | 96 | 195
  Maintenance Phase - Male | 0 | 0 | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Induction Phase: Number of Patients Showing Treatment Response
Description: Treatment response was adjudicated by a blinded clinical endpoints committee (CEC) and defined as: a) Decrease in proteinuria, defined as a decrease in the urine protein to creatinine ratio (UPCr) to <3 in subjects with baseline proteinuria ≥3 UPCr or a decrease in the UPCr by ≥50% in subjects with proteinuria <3 UPCr at Baseline, and b) Stabilization of serum creatinine or improvement. UPCr were derived from the 24 hour urine collection. Patients who did not show a treatment response at Week 24 or who withdrew earlier than Week 24 were considered non-responders.
Time Frame: 24 weeks
Population: Analysis population was intent to treat which comprised all subjects who were randomized into the study and had at least one post-baseline efficacy assessment.
Measure: Number; unit: participants
Groups:
- Intravenous Cyclophosphamide: Participants received monthly intravenous infusions of cyclophosphamide, 0.5 to 1.0 g per square meter of body surface area and concomitant treatment with corticosteroids for the 24 week Induction Phase.
- Mycophenolate Mofetil: Participants received oral mycophenolate mofetil (MMF) 1.5 g twice a day and concomitant corticosteroids for the 24-weeks of the Induction Phase.
Arm/Group | Intravenous Cyclophosphamide | Mycophenolate Mofetil
Number analyzed (Participants) | 185 | 185
participants
  Responder | 98 | 104
  Non-responder | 87 | 81
Statistical Analysis 1: Comparison: Intravenous Cyclophosphamide vs Mycophenolate Mofetil; Test type: Superiority or Other; p = 0.478, Regression, Logistic; Covariates included Treatment, Race, Geographical Region, and WHO Lupus Nephritis Class V and specified interaction terms

2. Primary Outcome: Maintenance Phase: Kaplan-Meier Estimates of Percentage of Participants Treatment Failure Free, by Time Interval
Description: Treatment Failure was adjudicated by a clinical endpoints committee and was defined as the time to the earliest occurrence of any one of the following: death, end stage renal disease, sustained doubling of serum creatinine, renal flare, or a requirement for rescue therapy for exacerbation or deterioration of Lupus nephritis. Kaplan-Meier survival curves were estimated from the observed time to treatment failure for each patient. The data presented are the percentage of participants who were treatment-failure free at each time interval as estimated by Kaplan-Meier.
Time Frame: From the start of the Maintenance Phase to Month 36
Population: Intent to treat analysis population which consisted of all subjects who were randomized to the maintenance phase of the study and had at least 1 maintenance efficacy assessment.
Measure: Number; unit: Percentage of participants
Groups:
- Mycophenolate Mofetil: Participants who responded to Induction Phase treatment received mycophenolate mofetil (MMF) 1.0 g orally twice a day, placebo to azathioprine orally once a day and corticosteroid for the 36 weeks Maintenance Phase.
- Azathioprine: Participants who responded to Induction Phase treatment received azathioprine (AZA) 2 mg/kg/day orally once a day, placebo to mycophenolate mofetil orally twice a day and corticosteroid for the 36 weeks Maintenance Phase.
Arm/Group | Mycophenolate Mofetil | Azathioprine
Number analyzed (Participants) | 116 | 111
Percentage of participants
  Start of Maintenance Phase to Month 3 | 98.2 | 97.2
  Month 3 to Month 6 | 93.7 | 89.3
  Month 6 to Month 9 | 89.9 | 86.2
  Month 9 to Month 12 | 86.0 | 83.0
  Month 12 to Month 15 | 86.0 | 77.5
  Month 15 to Month 18 | 84.9 | 74.1
  Month 18 to Month 21 | 84.9 | 70.7
  Month 21 to Month 24 | 83.9 | 68.3
  Month 24 to Month 27 | 82.8 | 67.1
  Month 27 to Month 30 | 82.8 | 65.9
  Month 30 to Month 33 | 81.7 | 63.4
  Month 33 to Month 36 | 81.7 | 58.6
Statistical Analysis 1: Comparison: Mycophenolate Mofetil vs Azathioprine; The difference in Kaplan-Meier survival curves between treatment groups (MMF-AZA) was assessed using a log-rank test, which is a non-parametric test to compare the survival distributions of two groups commonly used to analyze time-to-event endpoints; Test type: Superiority or Other; p = 0.003, Log Rank — Testing at the alpha=0.05 level was applied with no adjustments made for multiplicity

3. Secondary Outcome: Induction Phase: Number of Participants Achieving Complete Remission
Description: Number of participants achieving complete remission as defined by return to normal serum creatinine, proteinuria ≤500 mg/24 hours and an inactive urinary sediment (absence of red blood cells, white blood cells or cellular or granular casts) after 24 weeks.
Time Frame: 24 weeks
Population: Analysis population was intent to treat.
Measure: Number; unit: participants
Arm/Group | Intravenous Cyclophosphamide | Mycophenolate Mofetil
Number analyzed (Participants) | 185 | 185
participants
  Complete Remission - Yes | 15 | 16
  Complete Remission - No | 170 | 169

4. Secondary Outcome: Induction Phase: Change From Baseline to Week 24 in Serum Creatinine
Time Frame: Baseline, Week 24
Population: Analysis population was intent to treat. The analysis included only those patients for whom data was available at both time points, as indicated by "n".
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Intravenous Cyclophosphamide | Mycophenolate Mofetil
Number analyzed (Participants) | 185 | 185
µmol/L
  Baseline [n= 184, 185] | 92.7 (56.88) | 108.6 (97.21)
  Week 24 [n= 155, 151] | 83.5 (56.26) | 77.6 (35.08)
  Change from Baseline to Week 24 [n= 154, 151] | -5.1 (45.96) | -18.9 (59.03)

5. Secondary Outcome: Induction Phase: Change From Baseline to Week 24 in 24-hour Urine Protein
Description: 24-hour urine protein was measured at Baseline and Week 24.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Intravenous Cyclophosphamide | Mycophenolate Mofetil
Number analyzed (Participants) | 185 | 185
mg/day
  Baseline [n=180, 180] | 4451.4 (3506.59) | 4208.9 (3347.34)
  Week 24 [n= 150, 144] | 1831.6 (2413.84) | 1599.0 (2165.80)
  Change from Baseline to Week 24 [n= 146, 142] | -2513.7 (3223.68) | -2510.6 (3132.69)

6. Secondary Outcome: Induction Phase: Change From Baseline to Week 24 in Serum Albumin
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Intravenous Cyclophosphamide | Mycophenolate Mofetil
Number analyzed (Participants) | 185 | 185
g/L
  Baseline [n=184, 185] | 28.6 (6.98) | 30.5 (6.90)
  Week 24 [n=155, 151] | 38.3 (6.16) | 38.4 (5.50)
  Change from Baseline to Week 24 [n=154, 151] | 9.0 (6.77) | 7.5 (6.25)

7. Secondary Outcome: Induction Phase: Change in Renal British Isles Lupus Assessment Group (BILAG) Score
Description: BILAG indices provide a scoring system for the assessment of lupus disease activity in terms of the need for steroid treatment in 8 organs/systems. Eighty-six items were scored resulting in a classification of A (severe activity), B (moderate activity), C (mild activity), D (no current activity) and E (no activity ever observed) for each organ system. The BILAG individual system summaries were calculated by a program supplied by ADS-Limathon (Sheffield, UK).
  The score at baseline was compared to the score at the 24 week endpoint for each treatment group, reported here for the renal system.
Time Frame: Baseline, 24 weeks
Population: Analysis population was intent to treat. The endpoint was defined using the last observation carried forward approach. If no post-Baseline value was available, endpoint was considered missing.
Measure: Number; unit: Percentage of participants
Arm/Group | Intravenous Cyclophosphamide | Mycophenolate Mofetil
Number analyzed (Participants) | 181 | 181
Percentage of participants
  Shift from Baseline=A to 24 Week Endpoint=A | 27.1 | 17.1
  Shift from Baseline=A to 24 Week Endpoint=B | 34.8 | 39.2
  Shift from Baseline=A to 24 Week Endpoint=C | 24.9 | 33.1
  Shift from Baseline=A to 24 Week Endpoint=D | 9.4 | 5.5
  Shift from Baseline=B to 24 Week Endpoint=A | 0.0 | 0.0
  Shift from Baseline=B to 24 Week Endpoint=B | 1.1 | 1.7
  Shift from Baseline=B to 24 Week Endpoint=C | 1.7 | 2.2
  Shift from Baseline=B to 24 Week Endpoint=D | 0.0 | 1.1
  Shift from Baseline=C to 24 Week Endpoint=A | 0.0 | 0.0
  Shift from Baseline=C to 24 Week Endpoint=B | 0.6 | 0.0
  Shift from Baseline=C to 24 Week Endpoint=C | 0.0 | 0.0
  Shift from Baseline=C to 24 Week Endpoint=D | 0.0 | 0.0
  Shift from Baseline=D to 24 Week Endpoint=A | 0.0 | 0.0
  Shift from Baseline=D to 24 Week Endpoint=B | 0.0 | 0.0
  Shift from Baseline=D to 24 Week Endpoint=C | 0.6 | 0.0
  Shift from Baseline=D to 24 Week Endpoint=D | 0.0 | 0.0

8. Secondary Outcome: Induction Phase: Change From Baseline in Short-Form Health Survey (SF-36) Domain and Component Scores
Description: The SF-36 is a 36 item quality of life questionnaire. The short-form version has eleven questions that permit the participant to rate how they feel that particular day. The SF-36 consists of eight scaled scores and two component scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 score with the higher scores indicating better quality of life.
Time Frame: Baseline and 24 weeks
Population: This analysis population is intention to treat. The analysis included only those patients for whom data was available at both time points, as indicated by "n".
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Intravenous Cyclophosphamide | Mycophenolate Mofetil
Number analyzed (Participants) | 185 | 185
Scores on a scale
  Physical Component Summary [n=139, 137] | 6.4 (8.74) | 5.2 (8.60)
  Mental Component Summary [n=139, 137] | 5.7 (11.39) | 6.7 (11.45)
  Bodily Pain Score [n=141, 137] | 16.8 (25.85) | 13.4 (24.57)
  General Health Score [n=139, 137] | 11.5 (20.90) | 9.1 (19.49)
  Mental Health Score [n=141, 137] | 9.8 (19.47) | 9.3 (18.96)
  Physical functioning Score [n=141, 137] | 9.3 (24.63) | 11.6 (23.12)
  Role-Emotional Score [n=141, 137] | 18.4 (46.71) | 23.4 (44.90)
  Role-Physical Score [n=141, 137] | 34.0 (47.65) | 28.6 (48.18)
  Social Function Score [n=141, 137] | 18.2 (29.26) | 17.7 (28.06)
  Vitality Score [n=141, 137] | 11.6 (20.68) | 14.2 (23.30)

9. Secondary Outcome: Maintenance Phase: Events Contributing to the Primary Endpoint: Number of Deaths
Description: Treatment Failure was adjudicated by a clinical endpoints committee (CEC) and was defined as the time to the earliest occurrence of any one of the following: death, end stage renal disease, sustained doubling of serum creatinine, renal flare, or a requirement for rescue therapy for exacerbation or deterioration of Lupus nephritis (LN).
Time Frame: From the start of the Maintenance Phase to Month 36
Population: Maintenance Phase intent to treat population.
Measure: Number; unit: Deaths
Groups:
- Mycophenolate Mofetil (MMF): Mycophenolate mofetil (MMF) 1.0 g orally twice a day + Placebo to Azathioprine orally once a day + Corticosteroid for 36 months
- Azathioprine (AZA): Azathioprine (AZA) 2 mg/kg/day orally once a day + Placebo to MMF orally twice a day + Corticosteroid for 36 months.
Arm/Group | Mycophenolate Mofetil (MMF) | Azathioprine (AZA)
Number analyzed (Participants) | 116 | 111
Deaths | 0 | 1

10. Secondary Outcome: Maintenance Phase: Events Contributing to the Primary Endpoint: Number of Participants With End-stage Renal Disease (ESRD)
Description: Time to treatment failure, adjudicated by the Clinical Endpoints Committee (CEC), was defined as any 1 the following: death, ESRD, sustained doubling of serum creatinine, renal flare (proteinuric or nephritic), or requirement for rescue therapy to treat deterioration or exacerbation of Lupus nephritis. ESRD is defined as progression to chronic hemodialysis or renal transplant.
Time Frame: From the start of the Maintenance Phase to Month 36
Population: Maintenance Phase intent to treat population. The analysis includes all event data, regardless of whether or not the event was the earliest Clinical Endpoints Committee-adjudicated reason for treatment failure.
Measure: Number; unit: participants
Groups:
- Mycophenolate Mofetil (MMF): Mycophenolate mofetil (MMF) 1.0 g twice daily (BID) along with placebo matching AZA (2.0 mg/kg/day), plus corticosteroid, until 36 months of therapy.
- Azathioprine (AZA): Azathioprine (AZA) 2.0 mg/kg/day along with placebo matching MMF (1.0 g BID), plus corticosteroid for 36 months of therapy
Arm/Group | Mycophenolate Mofetil (MMF) | Azathioprine (AZA)
Number analyzed (Participants) | 116 | 111
participants | 0 | 3

11. Secondary Outcome: Maintenance Phase: Events Contributing to the Primary Endpoint: Number of Participants With Sustained Doubling of Serum Creatinine
Description: Sustained doubling of serum creatinine concentration is defined as the first serum creatinine value that is twice the mean of the lowest 2 values from screening to end of induction, as confirmed by a second serum creatinine value obtained at least 4 weeks after the initial doubling.
Time Frame: From the start of the Maintenance Phase to Month 36
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Azathioprine
Number analyzed (Participants) | 116 | 111
participants | 1 | 5

12. Secondary Outcome: Maintenance Phase: Events Contributing to the Primary Endpoint: Kaplan-Meier Estimates of Percentage of Participants Renal Flare Free, by Time Interval
Description: A proteinuric flare is defined as a doubling of the urine protein:creatinine ratio, and proteinuria ≥1 g/24 h in patients with urine protein ≤0.5 g/24 h at the end of the induction phase, or proteinuria ≥2 g/24 h if urine protein was >0.5 g/24 h at the end of the induction phase. A nephritic flare is defined as a 25% increase in serum creatinine accompanied by 1 or more of the following: (a) simultaneous doubling of the proteinuria reaching a minimum of 2 g/24 h (b) new/increased hematuria or (c) the appearance of cellular casts. All flares were adjudicated by a clinical endpoints committee.
Time Frame: From the start of the Maintenance Phase to Month 36
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Mycophenolate Mofetil | Azathioprine
Number analyzed (Participants) | 116 | 111
Percentage of participants
  Start of Maintenance Phase to Month 3 | 98.2 | 97.2
  Month 3 to Month 6 | 94.6 | 90.3
  Month 6 to Month 9 | 90.8 | 87.2
  Month 9 to Month 12 | 87.8 | 85.0
  Month 12 to Month 15 | 87.8 | 82.8
  Month 15 to Month 18 | 86.8 | 79.2
  Month 18 to Month 21 | 86.8 | 78.0
  Month 21 to Month 24 | 86.8 | 75.5
  Month 24 to Month 27 | 86.8 | 74.2
  Month 27 to Month 30 | 86.8 | 74.2
  Month 30 to Month 33 | 85.6 | 72.9
  Month 33 to Month 36 | 85.6 | 70.1

13. Secondary Outcome: Maintenance Phase: Events Contributing to the Primary Endpoint: Kaplan-Meier Estimates of Percentage of Participants Not Receiving Rescue Therapy
Description: The primary efficacy parameter was the time to treatment failure, adjudicated by the Clinical Endpoints Committee (CEC), defined as any of the following: death, end stage renal disease, sustained doubling of serum creatinine, renal flare, or requirement for rescue therapy to treat deterioration or exacerbation of Lupus nephritis. Kaplan-Meier survival curves were estimated from the observed time to rescue treatment for each patient. The data presented are the percentage of participants who were rescue treatment free at each time interval as estimated by Kaplan-Meier.
Time Frame: From the start of the Maintenance Phase to Month 36
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Mycophenolate Mofetil | Azathioprine
Number analyzed (Participants) | 116 | 111
Percentage of participants
  Start of Maintenance Phase to Month 3 | 100 | 99.1
  Month 3 to Month 6 | 98.2 | 95.1
  Month 6 to Month 9 | 97.2 | 93.0
  Month 9 to Month 12 | 94.2 | 91.9
  Month 12 to Month 15 | 94.2 | 88.4
  Month 15 to Month 18 | 94.2 | 87.1
  Month 18 to Month 21 | 93.1 | 83.1
  Month 21 to Month 24 | 91.9 | 83.1
  Month 24 to Month 27 | 90.8 | 81.7
  Month 27 to Month 30 | 90.8 | 80.3
  Month 30 to Month 33 | 90.8 | 78.8
  Month 33 to Month 36 | 90.8 | 75.9

14. Secondary Outcome: Maintenance Phase: Participants With Major Extra-renal Flare
Description: A major extra-renal flare is defined as a British Isles Lupus Assessment Group (BILAG) Score category A in one extrarenal organ or three organs with concurrent category B scores. BILAG indices provide a scoring system for the assessment of lupus disease activity in terms of the need for steroid treatment in 8 organs/systems. Eighty-six items were scored resulting in a classification of A (severe activity), B (moderate activity), C (mild activity), D (no current activity) and E (no activity ever observed) for each organ system.
Time Frame: From the start of the Maintenance Phase to Month 36
Population: Maintenance Phase intent to treat population.
Measure: Number; unit: participants
Arm/Group | Mycophenolate Mofetil | Azathioprine
Number analyzed (Participants) | 116 | 111
participants | 7 | 6

ADVERSE EVENTS:
Time Frame: AEs were monitored from the time of informed consent throughout the course of the study (up to 42 months).
Description: The induction and maintenance phases were analyzed separately. All safety analyses are based on the safety population.
Arm/Group | Induction Phase: Cyclophosphamide | Induction Phase: Mycophenolate Mofetil | Maintenance Phase: Mycophenolate Mofetil | Maintenance Phase: Azathioprine
Serious Adverse Events (participants affected / at risk) | 41/180 | 51/184 | 27/115 | 37/111
Other Adverse Events (participants affected / at risk) | 171/180 | 177/184 | 113/115 | 108/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Cyclophosphamide (N=180) | Induction Phase: Mycophenolate Mofetil (N=184) | Maintenance Phase: Mycophenolate Mofetil (N=115) | Maintenance Phase: Azathioprine (N=111)
Pneumonia (Infections and infestations) | 3 | 5 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 5 | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 2 | 0 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Subacute endocarditis (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 3 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 2 | 1 | 5
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 2 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Lupus encephalitis (Nervous system disorders) | 2 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 3 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 3 | 6
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0
Venous stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Biopsy kidney (Investigations) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 2
Peridiverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Genitourinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic hematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Superior sagittal sinus thrombosis (Nervous system disorders) | 0 | 0 | 0 | 1
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Peripheral ischemia (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Abnormal behavior (Psychiatric disorders) | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 0 | 2 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Phase: Cyclophosphamide (N=180) | Induction Phase: Mycophenolate Mofetil (N=184) | Maintenance Phase: Mycophenolate Mofetil (N=115) | Maintenance Phase: Azathioprine (N=111)
Nasopharyngitis (Infections and infestations) | 29 | 25 | 15 | 13
Upper respiratory tract infection (Infections and infestations) | 28 | 17 | 41 | 36
Herpes zoster (Infections and infestations) | 6 | 14 | 7 | 6
Urinary tract infection (Infections and infestations) | 17 | 19 | 20 | 27
Diarrhoea (Gastrointestinal disorders) | 23 | 52 | 22 | 20
Nausea (Gastrointestinal disorders) | 82 | 27 | 20 | 21
Vomiting (Gastrointestinal disorders) | 68 | 25 | 14 | 18
Abdominal pain (Gastrointestinal disorders) | 13 | 19 | 11 | 14
Abdominal pain upper (Gastrointestinal disorders) | 18 | 15 | 13 | 11
Constipation (Gastrointestinal disorders) | 9 | 12 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 10 | 3 | 7
Oedema peripheral (General disorders) | 30 | 35 | 8 | 7
Oedema (General disorders) | 17 | 11 | 0 | 0
Fatigue (General disorders) | 18 | 18 | 17 | 20
Asthenia (General disorders) | 15 | 9 | 6 | 6
Chest pain (General disorders) | 10 | 8 | 0 | 0
Pyrexia (General disorders) | 30 | 12 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 64 | 20 | 12 | 11
Rash (Skin and subcutaneous tissue disorders) | 21 | 19 | 15 | 14
Acne (Skin and subcutaneous tissue disorders) | 9 | 9 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 10 | 5 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 29 | 29 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 19 | 13 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 6 | 10 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 10 | 4 | 8 | 11
Headache (Nervous system disorders) | 47 | 38 | 25 | 27
Dizziness (Nervous system disorders) | 10 | 8 | 5 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 24 | 16 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 4 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 13 | 6 | 1
Anaemia (Blood and lymphatic system disorders) | 12 | 23 | 13 | 17
Leukopenia (Blood and lymphatic system disorders) | 38 | 11 | 26 | 40
Neutropenia (Blood and lymphatic system disorders) | 12 | 3 | 0 | 0
Hypertension (Vascular disorders) | 25 | 26 | 8 | 7
White blood cell count decreased (Investigations) | 16 | 5 | 0 | 0
Insomnia (Psychiatric disorders) | 11 | 10 | 11 | 3
Palpitations (Cardiac disorders) | 6 | 11 | 0 | 0
Tachycardia (Cardiac disorders) | 6 | 10 | 0 | 0
Cushingoid (Endocrine disorders) | 11 | 9 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 10 | 4
Pharyngitis (Infections and infestations) | 0 | 0 | 6 | 6
Bronchitis (Infections and infestations) | 0 | 0 | 14 | 7
Gastroenteritis (Infections and infestations) | 0 | 0 | 16 | 6
Influenza (Infections and infestations) | 0 | 0 | 13 | 14
Respiratory tract infection (Infections and infestations) | 0 | 0 | 7 | 3
Gastritis (Gastrointestinal disorders) | 0 | 0 | 11 | 7
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 8 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 5 | 9
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 7 | 11
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 8
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7 | 5
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 15
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 7
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 3 | 9
Lupus nephritis (Renal and urinary disorders) | 0 | 0 | 17 | 25
Proteinuria (Renal and urinary disorders) | 0 | 0 | 11 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 4 | 6
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 3 | 6

LIMITATIONS AND CAVEATS:
For many of the Maintenance Phase Outcomes, the total number of events precluded a meaningful time to event statistical analysis, therefore, only events numbers are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.